CLINICAL TRIAL: NCT03579173
Title: Determinants of Early Cystic Fibrosis Lung Disease
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Heather Nicole Muston, Assistant Professor of Clinical Pediatrics, Indiana University School of Medicine
Other Study IDs: 1712581512
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Cystic Fibrosis in Children
Keywords: Nutritional Status; Infant Pulmonary Function Testing; Lung Clearance Index; Multiple Breath Washout

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Nutrition and Infant PFT: To examine the relationship between nutritional status (weight-for-age (WFA) and weight-for-length (WFL)) at 6 months of age and lung function at 1-2 years of age in infants with CF.
  Interventions: Diagnostic Test: Infant PFT
- Nutrition and Lung Clearance Index: To examine the relationship between nutritional status (WFA and WFL) in infants with CF at 12 months of age and the lung clearance index (LCI) at 3-5 years of age.
  Interventions: Diagnostic Test: Lung Clearance Index
- Passive Tidal Breathing and Infant PFT: To delineate the relationship between passive tidal breathing lung function testing in infants with CF at 4-8 weeks of age and subsequent lung function at 6-12 months of age.
  Interventions: Diagnostic Test: Infant PFT; Diagnostic Test: Passive tidal breathing

INTERVENTIONS:
Diagnostic Test: Infant PFT — Assessed through the raised volume rapid thoracoabdominal compression technique and plethysmography
  Groups: Nutrition and Infant PFT; Passive Tidal Breathing and Infant PFT
Diagnostic Test: Lung Clearance Index — The Lung Clearance Index is derived from the Multiple Breath Washout test. It is the cumulative exhaled volume (the volume of gas needed to wash out resident gas mixture out of the lungs) divided by the FRC. The FRC is the amount of air left in the lungs after normal exhalation.
  Groups: Nutrition and Lung Clearance Index
Diagnostic Test: Passive tidal breathing — During quiet sleep, tidal breathing flow-volume curves are obtained. The tPEF/tE is calculated by taking the time it takes to reach peak expiratory flow divided by the total peak expiratory time.
  Groups: Passive Tidal Breathing and Infant PFT

SUMMARY:
The overall objective of this study is to determine the impact early nutritional and respiratory indices have on early CF lung disease. This knowledge will guide clinical management of infants with CF, who are now primarily diagnosed through newborn screening.

DETAILED DESCRIPTION:
The overall objective of this study is to determine the impact early nutritional and respiratory indices have on early CF lung disease. This knowledge will guide clinical management of infants with CF, who are now primarily diagnosed through newborn screening. We hypothesize that respiratory and nutritional indices during the first year of life are critical determinants of lung function in infants and preschoolers with CF.

Aim #1 - To examine the relationship between nutritional status (weight-for-age (WFA) and weight-for-length (WFL)) at 6 months of age and lung function at 1-2 years of age in infants with CF.

Hypothesis: Infants with CF with poor nutritional status at 6 months of age will have worse lung function, as assessed through the raised volume rapid thoracoabdominal compression technique and plethysmography, compared to those with better nutritional indices, defined as improved weight-for-age and weight-for-length.

Aim #2 - To examine the relationship between nutritional status (WFA and WFL) in infants with CF at 12 months of age and the lung clearance index (LCI) at 3-5 years of age.

Hypothesis: Infants with CF with poor nutritional indices at 12 months of age will have a higher (worse) LCI at 3-5 years of age compared to those with better nutritional status.

Aim #3 - To delineate the relationship between passive tidal breathing lung function testing in infants with CF at 4-8 weeks of age and subsequent lung function at 6-12 months of age.

Hypothesis: Abnormalities in passive tidal breathing lung function testing will be associated with abnormal infant pulmonary function testing obtained via the raised volume rapid thoracoabdominal compression technique and plethysmography at 6-12 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by a parent or legal guardian
* A confirmed diagnosis of CF by newborn screening and either a documented sweat chloride of at least 60 mEq/L by quantitative pilocarpine iontophoresis or a genotype with two CF-causing mutations
* One month to five years of age.

Exclusion Criteria:

* Chronic lung disease not due to CF
* Contraindications to sedation, including structural abnormalities of the upper airway or chest wall and severe gastroesophageal reflux
* Gestational age < 36 weeks

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants and preschoolers with cystic fibrosis diagnosed by newborn screen.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Lung function | 24 months
  Forced expiratory volume in 0.5 seconds

SECONDARY OUTCOMES:
Lung function - FRC | 24 months
  Functional Residual Capacity
Lung function - MBW | 24 months
  Multiple breath washout result

CONTACTS AND LOCATIONS:
Overall Officials: Heather Muston, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No